CLINICAL TRIAL: NCT07191717
Title: Phase II Minimal Residual Disease Study of Selective Estrogen Receptor Degrader Imlunestrant With Cyclin-Dependent Kinase (CDK) 4/6 Inhibitor Abemaciclib in Patients With ER+ Breast Cancer (MIRI)
Brief Title: Imlunestrant and Abemaciclib for the Treatment of Estrogen Receptor Positive Breast Cancer in Patients With Minimal Residual Disease, MIRI Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-0200; NCI-2025-06030 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-09

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Invasive Breast Carcinoma; Localized Estrogen Receptor-Positive Breast Carcinoma; Localized Human Epidermal Growth Factor Receptor (HER2)-Negative Breast Carcinoma
MeSH Terms: interventions — abemaciclib; Specimen Handling; Imlunestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (abemaciclib, imlunestrant) (Experimental): Patients receive abemaciclib PO BID and imlunestrant PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection throughout the study. Patients may also undergo radiological scans per the discretion of the treating physician throughout the study.
  Interventions: Drug: Abemaciclib; Procedure: Biospecimen Collection; Drug: Imlunestrant; Other: Questionnaire Administration; Procedure: Radiologic Imaging Procedure

INTERVENTIONS:
Drug: Abemaciclib — Given PO
  Other Names: LY 2835219; LY-2835219; LY2835219; Verzenio
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Imlunestrant — Given PO
  Other Names: LY 3484356; LY-3484356; LY3484356; Selective Estrogen Receptor Degrader LY3484356; SERD LY3484356
Other: Questionnaire Administration — Ancillary studies
Procedure: Radiologic Imaging Procedure — Undergo radiologic scans

SUMMARY:
This phase II trial studies how well imlunestrant and abemaciclib work in treating patients with estrogen receptor positive (ER+) breast cancer who have tumor remaining in the blood following treatment (minimal residual disease). Estrogen can cause the growth of breast cancer cells. Imlunestrant lowers the amount of estrogen made by the body. This may help stop the growth of tumor cells that need estrogen to grow. Abemaciclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Imlunestrant and abemaciclib may be effective in treating patients with ER+ breast cancer who have minimal residual disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the rate of circulating tumor deoxyribonucleic acid (ctDNA) clearance after 12 cycles of adjuvant imlunestrant and abemaciclib.

SECONDARY OBJECTIVES:

I. To investigate the safety and tolerability of 12 cycles of adjuvant imlunestrant and abemaciclib.

II. To assess the rate of ctDNA re-emergence in the 12 cycles following treatment on imlunestrant and abemaciclib.

III. To evaluate the 1-year distant recurrence-free survival (DRFS), defined as the time from enrollment to evidence of distant disease recurrence or death due to any cause.

EXPLORATORY OBJECTIVE:

I. To assess potential predictive biomarkers of response to imlunestrant and abemaciclib.

OUTLINE:

Patients receive abemaciclib orally (PO) twice daily (BID) and imlunestrant PO once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection throughout the study. Patients may also undergo radiological scans per the discretion of the treating physician throughout the study.

After completion of study treatment, patients are followed up at 30 days and then every 4 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have localized ER+ (≥ 10% on surgical pathology), HER2 negative, any grade, invasive breast cancer. Pathological stage (from time of surgery, including patients who received neoadjuvant therapy) I - III by American Joint Committee on Cancer (AJCC) 8th edition staging

  * Note: Invasive breast cancer must be ER+ in ≥ 10% of the cells and HER2 negative (immunohistochemistry [IHC] 0 or 1+ and/or fluorescence in situ hybridization [FISH] negative with a ratio < 2) by American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines. For Immunohistochemistry (IHC) 2+, the tumor must be FISH negative with a ratio < 2. ER, progesterone receptor (PR) and HER2 measurements should be performed according to institutional (local) guidelines, in a Clinical Laboratory Improvement Act (CLIA)-approved setting
* Detectable ctDNA in a CLIA-certified lab (separate pre-screening consent available) within the past six months. Participants must have no clinical or radiographic evidence of recurrence as determined by the treating investigator
* Confirmation of adequate archival tissue (either initial biopsy or surgical specimen) (15-20 unstained slides cut at 5 µm or 1 block) required before study entry. If adequate surgical tissue is available, this is preferred. Otherwise tissue from diagnostic biopsy is acceptable. If adequate tissue not available, principal investigator (PI) approval is required prior to study entry
* No prior history of other malignancies within past 5 years (besides breast cancer as per inclusion #1). Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: ductal carcinoma in situ of the breast, cervical cancer in situ, melanoma in situ, and basal cell or squamous cell carcinoma of the skin. No concurrent malignancy or other serious medical condition as deemed by the investigator
* Participants may or may not have received (neo)adjuvant chemotherapy and/or biological therapy at the time of screening, with no more than grade 1 residual toxicity (except ≤ grade 2 neuropathy or ≤ grade 2 alopecia)
* Participants may or may not have received adjuvant radiotherapy, with no more than grade 1 residual toxicity
* Pre- and postmenopausal women and men are eligible. Premenopausal women must have a negative serum pregnancy test at time of screening

  * Pregnancy testing does not need to be pursued in female patients who are:

    * Age ≥ 60 years; OR
    * Age < 60 with intact uterus AND amenorrhea for 12 consecutive months or more AND estrogen (estradiol) levels within postmenopausal range
    * OR status-post bilateral oophorectomy, total hysterectomy, or bilateral tubal ligation
* Must be ≥ 18 years of age
* History of CDK 4/6 inhibitor is permitted provided the last dose was more than 6 months ago (from consent date)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (Karnofsky ≥ 70%)
* Patients must currently be on endocrine therapy in the adjuvant setting and must have received (neo) adjuvant endocrine therapy for at least 24 months (cumulative duration)
* Ability to understand and the willingness to sign a written informed consent document. Patient must sign the informed consent (ICF) prior to any screening procedures being performed and is able to comply with protocol requirements
* Participants must currently be receiving adjuvant endocrine therapy and have been on adjuvant endocrine therapy for at least 2 years. Adjuvant endocrine therapy can be either tamoxifen or aromatase inhibitor (AI), i.e prior use of any AI, including letrozole, anastrozole or exemestane, or tamoxifen is allowed. Concurrent gonadotrophin releasing hormone (GNRH) agonist is required with AI in pre - and/or peri-menopausal patients and men
* Absolute neutrophil count ≥ 1.5 × 10^9/L
* Platelets ≥ 100 × 10^9/L
* Hemoglobin ≥ 9.0 g/dL
* Serum creatinine < 1.5 mg/dL OR creatinine clearance ≥ 50 mL/min
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x institutional upper limit of normal (ULN)
* Total bilirubin < institutional 1.5 times ULN; or total bilirubin ≤ 3.0 x institutional ULN. Patients with Gilbert's Syndrome with a total bilirubin ≤ 2.0 times ULN and direct bilirubin within normal limits are permitted
* The patient is able to swallow oral medications

Exclusion Criteria:

* Participants with metastatic disease (including contralateral axillary lymph nodes) or inflammatory breast cancer. Of note, if a patient had locally advanced breast cancer leading to inflammation, this would not exclude the patient on the grounds of inflammatory carcinoma
* Participants who have had CDK 4/6 inhibitor therapy within the past 6 months. Use of prior CDK 4/6 inhibitor with last dose more than 6 months ago is permitted
* Participants who are receiving any other anti-cancer investigational agents. Participation in other observational studies is permitted
* History of other malignancies within past 5 years, except ductal carcinoma in situ of the breast, cervical cancer in situ, melanoma in situ, and basal cell or squamous cell carcinoma of the skin. No concurrent malignancy or other serious medical condition as deemed by the investigator
* Herbal products and supplements will generally not be allowed, but specific supplements (such as cannabidiol [CBD] oil) can be considered on a case-by-case basis by Overall PI
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment (e.g. estimated creatinine clearance < 30ml/min), unstable angina pectoris, cardiac arrhythmia, a preexisting chronic condition resulting in baseline grade 2 or higher diarrhea, or psychiatric illness/social situations that would limit compliance with study requirements. Patients with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, stomach resection, or small bowel resection) are ineligible. Patient with active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]). Screening for HIV and hepatitis is not required for enrollment
* The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest
* A history of venous thromboembolism (VTE): deep vein thrombus or pulmonary embolism. An exception can be made for patients with a history of an uncomplicated venous catheter-related occlusion. The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest
* History of hypersensitivity to imlunestrant, abemaciclib or any of the components in either medication
* HIV-positive participants not on antiretroviral therapy are at increased risk of lethal infections when treated with marrow-suppressive therapy and should not be enrolled until their HIV is managed. If the HIV is well controlled, participants may participate in this study
* Pregnant women are excluded from this study because embryo-fetal toxicity is a potential side effect of abemaciclib and imlunestrant. For this reason, women of child-bearing potential (WOCBP) and men must agree to use highly effective contraception prior to study entry, for the duration of treatment, and for at least 3 months after the completion of treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Prior to study enrollment, WOCBP must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential. All WOCBP must have a negative serum pregnancy test within 72 hours prior to receiving the first dose of the investigational agent(s). Registration may occur prior to this pregnancy test. If the pregnancy test is positive, the patient must not receive protocol treatment and must not continue in the study. WOCBP is defined as follows:

  * Any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or a bilateral oophorectomy) OR
  * Any female who is not postmenopausal defined as:

    * Age ≥ 60 years; OR
    * Age < 60 with intact uterus AND amenorrhea for 12 consecutive months or more AND estrogen (estradiol) levels within postmenopausal range; OR
    * Status-post bilateral oophorectomy, total hysterectomy, or bilateral tubal ligation
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception throughout the study and for 12 weeks after study drug discontinuation. Women are considered post-menopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of childbearing potential. Highly effective contraception methods include:

  * Total abstinence when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Use of non-estrogen oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception
  * Use of luteinizing hormone-releasing hormone (LHRH) agonist with estrogen level in post-menopausal range and one form of barrier method contraception
* Women who are lactating. Advise lactating women to not breastfeed during treatment and for 1 week after last dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2030-04-30 (Estimated); Study Completion 2031-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of circulating tumor deoxyribonucleic acid (ctDNA) clearance | After 12 cycles (Cycle length = 28 days)
  Clearance of ctDNA is defined as having undetectable plasma ctDNA after completion of 12 cycles of adjuvant imlunestrant and abemaciclib. The rate of ctDNA clearance will be calculated as the percentage of all enrolled patients that have undetectable plasma after completion of adjuvant imlunestrant and abemaciclib (12 cycles or sooner if trial therapy is discontinued), and its Wilson 95% confidence interval will be reported.

SECONDARY OUTCOMES:
Rate of ctDNA re-emergence | Up to 1 year after treatment
  Of participants with ctDNA clearance, rate of re-emergence of ctDNA (development of detectable ctDNA after previous ctDNA clearance) in the 12 cycles following treatment will be calculated. The time from discontinuation of protocol therapy to ctDNA re-emergence will be estimated using the Kaplan-Meier method.
Distant recurrence-free survival | From enrollment to evidence of distant disease recurrence or death due to any cause, assessed up to 1 year
  Will be estimated based on Kaplan-Meier method. Events will be defined as having clinical or radiographic evidence of distant metastatic recurrence or death due to any cause. Participants alive without distant disease recurrence will be censored at date of last evaluation. The distant recurrence will be determined by the treating investigator based on routine clinical evaluation and/or imaging, as part of standard follow-up. If recurrence is suspected, it will be confirmed by pathological confirmation to document carcinoma, as per as per National Comprehensive Cancer Network guidelines.
Incidence of adverse events | Up to 30 days after the last dose of study treatment
  Safety and tolerability will be determined by the investigator based on Common Terminology Criteria for Adverse Events version 5. The frequency and severity of adverse events will be summarized, and the proportion of patients who discontinue the treatment due to toxicity (and a Wilson 95% confidence interval) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Marla Lipsyc-Sharf, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States